CLINICAL TRIAL: NCT06990685
Title: Effect of Salidroside on Pregnancy Outcomes in High Childbearing Age Patients in Viro Fertilization: an Open-label Randomized Controlled Trial
Brief Title: Effect of Salidroside on Pregnancy Outcomes in High Childbearing Age Patients in Viro Fertilization
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Linlin Cui, Professor, The Second Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYLL2025357
Record Dates: First submitted 2025-04-21; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Salidroside; Randomized Controlled Trial; In Vitro Fertilization; Assisted Reproductive Technology
MeSH Terms: interventions — rhodioloside

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Long protocol, short protocol, or antagonist protocol et al.
- Experimental Group (Experimental): In the salidroside group, oral administration of rhodiola capsules (Xizang Gaoyuan 'an Biotechnology Development Co., LTD.) was started on the day of entering the COS cycle, once a day, 2 pills at a time, and the drug was stopped on the trigger day.
  Interventions: Drug: Salidroside

INTERVENTIONS:
Drug: Salidroside — In the salidroside group, oral administration of rhodiola capsules (Xizang Gaoyuan 'an Biotechnology Development Co., LTD.) was started on the day of entering the COS cycle, once a day, 2 pills at a time, and the drug was stopped on the trigger day.
  Arms: Experimental Group

SUMMARY:
With the decreasing of birth rate and population in our country, population problem has become a long-term and strategic problem. In addition to the decrease in the number of women of childbearing age and the impact of unmarried women, the increase in the incidence of reproductive disorders and the delay of marriage and childbearing are also important factors leading to the continuous decline of the birth population in China. Among them, ovarian aging is a key factor causing female fertility difficulties. Therefore, establishing an effective prevention and treatment strategy for ovarian aging is of great significance for improving female reproductive health and serving the national population strategy. Recently, several supplements have been found to promote folliculogenesis and improve oocyte quality. However, to date, there is no approved therapeutic agent for the treatment of ovarian aging. Therefore, it is urgent to develop effective strategies for the prevention and treatment of ovarian aging.

Salidroside is the main active component of Chinese medicine Rhodiola, and its content is highest in the root of rhodiola, which is also the main medicinal part. The main efficacy of salidroside in traditional Chinese medicine is to benefit qi, promote blood circulation, unblock pulse and relieve asthma. At the same time, in basic research, more and more experiments have shown that salidroside has a variety of pharmacological properties, including anti-hypoxia, anti-fatigue and anti-aging effects, anti-cancer, anti-inflammatory, anti-oxidation, antiviral and so on. These pharmacological effects suggest that salidroside may be an effective drug for the prevention and treatment of atherosclerosis, Parkinson's disease, Alzheimer's disease, pneumonia and other diseases. In terms of aging, it has been confirmed that salidroside supplementation can prolong the life span of pseudogill oryzias zhan and rescue premature aging of human skin fibroblasts, etc., which further confirms.

The aim of this study is to investigate the efficacy of salidroside as an adjuvant drug in improving the pregnancy outcomes of fresh embryo transfer in high childbearing age patients with poor ovarian response by comparing the pregnancy outcomes of fresh embryo transfer between salidroside group and blank control group. This pragmatic clinical study is expected to improve pregnancy outcomes of fresh embryo transfer cycles in women of advanced childbearing age with poor ovarian response.

DETAILED DESCRIPTION:
With the continuous decline in China's birth rate and number of births in recent years, the population issue has become a long-term and strategic issue in China. In addition to the impact of the decrease in the number of women of childbearing age and the non-marriage, the increase in the incidence of reproductive disorders and the postponement of the age of marriage and childbearing are also important factors leading to the continuous decline in the number of births in China. Among them, ovarian aging is a key factor causing fertility difficulties in women. Therefore, it is of great significance to establish an effective ovarian aging prevention and treatment strategy to improve women's reproductive health and serve the national population strategy. Recently, studies have found that a variety of supplements can promote follicular genesis and improve oocyte quality. However, to date, there are no approved effective treatments for ovarian aging. Therefore, it is urgent to develop effective strategies for the prevention and treatment of ovarian aging. Salidroside is the most active ingredient of Rhodiola rosea in traditional Chinese medicine, and has the highest content in the root of Rhodiola rosea, which is also the main medicinal site. The main effects of salidroside in traditional Chinese medicine are to invigorate qi and blood, and to relieve asthma. At the same time, in basic research, more and more experiments have shown that salidroside has a variety of pharmacological properties, including anti-hypoxia, anti-fatigue and anti-aging effects, anti-cancer effects, anti-inflammatory effects, antioxidant effects, antiviral effects, etc. These pharmacological effects suggest that salidroside may be an effective drug for the prevention and treatment of atherosclerosis, Parkinson's disease, Alzheimer's disease, pneumonia and other diseases. In terms of aging, it has been confirmed that supplementation of salidroside can prolong the life of Pseudogill medaka and save the premature aging of human skin fibroblasts, which further confirms the anti-aging effect and potential application value of salidroside. In the process of clinical assisted reproduction, the proportion of elderly women has been increasing in recent years; Due to the significant decline of female ovarian function in middle age, the success rate of assisted reproduction in elderly women has always been at a low level. However, whether in animal model studies or in human tissue sections, it is generally believed that there are still a large number of follicles in the ovaries of middle-aged females or females that are sufficient to support reproductive activities, but because the physiological reasons for the decline of ovarian function in middle-aged women are unknown, the contradiction of abundant follicles but declining ovarian function in middle-aged women cannot be overcome.Recently, Zhang Hua's team in China used high-resolution ovarian organ imaging technology combined with genetically modified animal models, single-cell omics and drug screening to reveal that the ovaries have specific vascular degeneration in middle age, which leads to a decrease in ovarian blood supply, stunted follicle development, and ultimately a decline in fertility. Mechanistic studies have confirmed that ovarian vascular endothelial aging is the cause of ovarian vascular degeneration in middle age. Based on the above findings, through the screening of a large number of natural products, it was found that in vitro treatment of salidroside can improve the regeneration ability of follicular blood vessels without affecting the development of follicles. Continuous injection of salidroside in vivo can significantly improve the ability of ovarian angiogenesis in elderly mice, improve ovarian blood supply, and then promote follicle development, increase the quantity and quality of ovulation in advanced mice, and increase the number of births in elderly mice. The safety evaluation proved that salidroside treatment had no effect on the blood vessels of heart, kidney, liver and other organs, and long-term (12 months) monitoring showed that there was no abnormal organ development and tumor production in mice after salidroside treatment. Other teams, using different in vitro and in vivo models, have also found that salidroside supplementation can improve oocyte quality in mice or pigs. On the one hand, the addition of salidroside to oocytes cultured in vitro can improve the maturation, fertilization and development ability of oocytes of childbearing age by maintaining normal spindle/chromosome structure and mitochondrial function, including improving oocyte spindle/chromosome arrangement, mitochondrial and cortical particle distribution, mitochondrial membrane potential, and reducing reactive oxygen species. On the other hand, it can also improve the oocyte quality of reproductive elderly mice by enhancing mitophagy, including improving their oocyte genesis, maturation, fertilization and embryonic development potential. The above studies provide a solid theoretical basis for salidroside to improve the quality of female oocytes. In summary, salidroside can improve oocyte quality and fertility through a variety of mechanisms. However, current research is still limited to animal experiments, and in-depth clinical evidence is lacking. Therefore, it is necessary to further explore the effect of salidroside on ovarian function, promote the clinical transformation of basic research, and serve the national population strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥35 and < 40 years old
2. For the first or second cycle of IVF, ICSI or IVF with donor sperm
3. According to the 2016 Poseton criteria for poor prognosis: the number of oocytes obtained in the previous routine ovulation induction protocol was 1-9, or AFC < 5 or AMH < 1.2ng/ml (measured within the past half year) in both ovaries.

Exclusion Criteria:

1. Patients with coagulation disorders
2. Patients with previous abnormal uterine bleeding
3. Combined with hydrosalpinx confirmed by B-ultrasound and HSG
4. Uterine malformation (unicornuate uterus, septate uterus) or history of intrauterine adhesions
5. Patients with previous spontaneous abortion ≥3 times
6. Patients with contraindications to assisted reproductive technology or pregnancy
7. Previous or current oral medication containing salidroside
8. The controlled ovarian stimulation protocol included PPOS protocol, luteal phase ovulation induction protocol, and continuous stimulation protocol

Ages: 35 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 370 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of continuous pregnancy cycles divided by the number of frozen embryo transfer cycles

SECONDARY OUTCOMES:
Clinical pregnancy rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of clinical pregnancy cycles divided by the number of transplantation cycles
Biochemical pregnancy rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of biochemical pregnancy cycles divided by the number of transplantation cycles
Live birth rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of live birth cycles divided by the number of transplantation cycles
Embryo implantation rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The ratio of the number of gestational sacs observed by ultrasound to the number of transplanted embryos
Early abortion rate | from transplantation to abortion (assessed up to 12 weeks of gestation)
  The ratio of the number of spontaneous abortion cycles to the number of clinical pregnancy cycles within 12 weeks of gestation
Ectopic pregnancy | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The embryo implants and grows and develops anywhere other than the uterine cavity
Pregnancy loss | from transplantation to abortion (assessed up to 28 weeks of gestation)
  Natural termination of clinical pregnancy or therapeutic induction of labor before 28 weeks of gestation
Stillbirth | from transplantation to delivery (assessed up to 40 weeks of gestation)
  A baby without vital signs is delivered at 28 weeks or more of gestation
Preterm birth | from transplantation to delivery (assessed up to 37 weeks of gestation)
  Delivery before 37 weeks of gestation
Gestational diabetes mellitus | from transplantation to delivery (assessed up to 40 weeks of gestation)
  Abnormalities of glucose metabolism of different degrees that first occur and are discovered during pregnancy
Preeclampsia | from transplantation to delivery (assessed up to 40 weeks of gestation)
  After 20 weeks of gestation, if a pregnant woman has a systolic blood pressure of ≥140 mmHg and/or a diastolic blood pressure of ≥90 mmHg, accompanied by any one of the following: urine protein quantification ≥0.3 g/24 h, or the urine protein/creatinine ratio ≥0.3, or random urine protein ≥(+)(the examination method when protein quantification is not performed unconditionally); There is no proteinuria but any one of the following organs or systems is involved: important organs such as the heart, lungs, liver, and kidneys, or abnormal changes in the blood system, digestive system, and nervous system, or the placenta and fetus are involved, etc.
Hypertension in Pregnancy | from transplantation to delivery (assessed up to 40 weeks of gestation)
  Hypertension first occurred after 20 weeks of pregnancy, with a systolic blood pressure of ≥140 mmHg (1 mmHg=0.133 kPa) and/or a diastolic blood pressure of ≥90 mmHg; The urine protein test was negative
Premature rupture of membranes | from transplantation to delivery (assessed up to 40 weeks of gestation)
  It refers to the spontaneous rupture of the fetal membranes before labor. According to the gestational age at which it occurs, it is divided into full-term fetal membranes and preterm premature rupture of fetal membranes
Placenta previa | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The lower edge of the placenta is adjacent to or covers the internal OS of the cervix
Placental abruption | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The placenta in its normal position partially or completely separates from the uterine wall before the fetus is delivered
Postpartum Hemorrhage | Within 24 hours after childbirth
  Within 24 hours after the delivery of the fetus, the amount of blood loss in parturients with vaginal delivery is ≥500 ml, the amount of blood loss in parturients with cesarean section is ≥ 1,000 ml, or there are symptoms or signs of hypovolume after blood loss
Neonatal death | Within 28 days after birth
  Infants with vital signs at birth die within 28 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Linlin Cui, M.D., Ph.D., Study Chair — The Second Hospital of Shandong University, China
Locations (1):
- The Second Hospital of Shandong University,, Jinan, Shandong, China